CLINICAL TRIAL: NCT05612698
Title: Efficacy of Different Modalities and Frequencies of Physical Exercise on Glucose Control in People With Prediabetes (Glycex Randomised Trial)
Brief Title: Efficacy of Physical Exercise on Glucose Control in People With Prediabetes
Acronym: GLYCEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Principal Investigator, Josep1, Full time teacher and researcher, University of the Balearic Islands
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GH2022/05
Record Dates: First submitted 2022-10-28; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: PreDiabetes
Keywords: prediabetes; aerobic training; resistance training; High intensive interval training
MeSH Terms: conditions — Prediabetic State | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The GLYCEX study (GLYcaemic Control with EXercise) is a randomised, parallel, phase II clinical trial with three active arms and a control group, with a duration of 15 weeks in each phase. Control group will receive general recommendations of PA, based on WHO recommendations, and after 15 weeks. Baseline evaluations will be repeated 15 weeks.
  Study interventions were reported using the Template for Intervention Description and Replication (TIDieR) as reference. The present protocol was elaborated following the Standard Protocol Items: Recommendations for Intervention Trials (SPIRIT) 2013 State-ment. Reporting of the study will follow the CONSORT statement recommendations on RCTs.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The sample size has been calculated to detect significant differences in FPG of at least 2 mg/dl and considering a standard destination of 2 mg/dl in any of the three modalities and a dropout rate of 10%, so 30 subjects will be needed in each group, with a sample of 90 participants. Furthermore, a control group (30 patients) will be added to evaluate the effect of any type of monitored exercise in these patients versus usual clinical practice. Randomization will be done by permuted blocks of 8 in a 1:1:1:1 ratio and participants will be stratified by gender, age and obesity using the open-source Oxford Minimization and Randomization (OxMaR) program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic training (Experimental): Aerobic Training intervention (AT): Perform 50 minutes/day, 3 days/week, totalling 150 min/week at moderate intensity, as recommended by WHO, in a range of 65-75% HRMax.
  Interventions: Behavioral: Aerobic training
- Aerobic training + resistance training (Experimental): Aerobic Training plus Resistance Training intervention (AT+RT): Perform 50 minutes/day, 3 days/week, starting with 50% of 1-repetition maximum (1-RM) and follow a progression of increasing loads up to 75% of 1-RM for optimal gains in strength and insulin action.
  Interventions: Behavioral: Aerobic training plus resistance training
- High Intensive Interval Training intervention (Experimental): High Intensive Interval Training intervention (HIIT): To be considered high intensive the heart rate needs to be above ≥85%. Perform 25 minutes/day, 3 days/week, totalling 75 min/week at a vigorous intensity, as recommended by WHO.
  Interventions: Behavioral: High intensive interval training
- Control (No Intervention): Participants in the control group will receive written standard PA recommendations in this phase.

INTERVENTIONS:
Behavioral: Aerobic training — Supervised Aerobic Training intervention (AT): Perform 50 minutes/day, 3 days/week, totalling 150 min/week at moderate intensity, as recommended by WHO, in a range of 65-75% HRMax. Due to any form of aerobic exercise involving large muscle groups and causes sustained increases in HR is likely to be beneficial, the type of aerobic exercise will be agreed with each group of patients, varying from 4 to 8 people. There will be a choice of ex-ercises and participants will be able to choose a combination of up to 2 different exercises. The participants' choice of the type of activity to be performed is expected to encourage greater adherence. The range of exercises will be brisk walking or running, swimming, and/or aerobic dancing.
  Arms: Aerobic training
Behavioral: Aerobic training plus resistance training — Supervised Aerobic Training plus Resistance Training intervention (AT+RT): Perform 50 minutes/day, 3 days/week, starting with 50% of 1-repetition maximum (1-RM) and follow a progression of increasing loads up to 75% of 1-RM for optimal gains in strength and insulin action. In each session, between 5 and 10 exercises will be worked on, per-forming 10-15 repetitions, and progressing to 8-10 lifting as the weight increases, involving the major muscle groups from the core, lower body and upper body. In all sessions there will be a 3-minute warm-up at the beginning of the session and a 2-minute cool-down at the end of the session.
  Arms: Aerobic training + resistance training
Behavioral: High intensive interval training — Supervised High Intensive Interval Training intervention (HIIT): To be considered high intensive the heart rate needs to be above ≥85%. Perform 25 minutes/day, 3 days/week, totalling 75 min/week at a vigorous intensity, as recommended by WHO. Starting with 4 intervals lasting 1 minute keeping in a range of 85-90% HRMax, separated by 1 minute of low intensity activity (no static) (4 × 1 min intervals.) A progression will be followed by increasing the number of circuits, up to 10 (10 × 1 min intervals) [25, 78, 79]. In all sessions there will be a 3-minute warm-up at the beginning of the session and a 2-minute cool-down at the end of the session. Although the target popula-tion is a sedentary population, we expect the HIIT approach, despite being high intensity, to be well received, due to its growing popularity, as demonstrated by a study in which 62% of inactive participants preferred HIIT to other types of exercise.
  Arms: High Intensive Interval Training intervention

SUMMARY:
To assess the efficacy of different modalities and frequencies of physical exercise on glycaemic control in adults with prediabetes. Methods: four-arm, parallel, randomised, controlled, clinical trial, with a total of 120 participants. A total of 90 participants will be randomized in three arms: 1) aerobic exercise, 2) aerobic exercise combined with resistance, and 3) high-intensity intervallic exercise. Moreover, a control group (n=30) will be included to evaluate the effect of any type of intervention versus no intervention. Data collection will be performed at baseline and 15-week of follow-up. Socio-demographic data, medication, comorbidity, blood biochemical parameters, blood pressure, anthropometric measurements, body composition, physical activity, sedentary lifestyle, diet, smoking, alcohol consumption, quality of life and sleep questionnaires will be collected. The main dependent variable will be the decrease of fasting plasma glucose. Moreover, a subsample of participants (n=40) will were an accelerometer and a continuous glycaemia monitoring during 7 days, in 2 time points. The impact of the interventions on health will be also evaluated through gene expression analysis in peripheral blood cells, widely used in clinical diagnosis in the same subsample. Discussion: The results of this study will contribute to improving physical exercise prescriptions for diabetes prevention, as well as a better understanding of the response of glucose mechanisms to physical exercise in a population with prediabetes. Increasing glycaemic control in people with prediabetes through physical exercise offers an opportunity to prevent diabetes and reduce associated comorbidities and health costs.

DETAILED DESCRIPTION:
Principal Aim. The main aim of the preset study is to compare the efficacy of 3 modalities of physical exercise on fasting plasma glucose in adults with prediabetes.

Secondary Aim. The secondary aims are to evaluate the effect of different physical exercise modalities on the following variables: glycaemic variability measured continuously (24h), normalization of glycaemic values (reversal), body mass index (BMI), body composition (percentage and grams of total fat mass and muscle mass; visceral adipose tissue (VAT) waist circumference, lipid profile, inflammation markers, blood pressure and sleep duration and quality; transcriptomic markers of metabolic health assessed in peripheral blood cells (PBC).

Design:

The GLYCEX study (GLYcaemic Control with EXercise) is a randomised, parallel, phase II clinical trial with four arms and a duration of 15 weeks. The intervention groups will receive an exercise intervention for 15 weeks, and control group will receive general recommendations of PA, based on world health organization (WHO) recommendations.

Study interventions were reported using the Template for Intervention Description and Replication (TIDieR). The present protocol was elaborated following the Standard Protocol Items: Recommendations for Intervention Trials (SPIRIT) 2013 State-ment. Reporting of the study will follow the CONSORT statement recommendations on RCTs.

Participants' identification and recruitment will be carried out at different primary care centres that formally agreed to participate in this phase, and through posters distributed at different points of interest: hospitals, universities, primary care centers, patient associations, etc. Likewise, it will also be disseminated through social networks, such as Twitter. Interested patients will receive the information sheet, sign the written informed consent and eligibility criteria will be verified.

Inclusion criteria: Adults aged 18-65 years, with overweight (BMI >25 and <35 Kg/m2), inactive (<150 min PA/week) and with prediabetes (fasting blood glucose 100-126 mg/dl) from primary care services in Mallorca, and who have signed the informed consent will be included.

Exclusion criteria: People with uncontrolled hypertension, diagnosis of type 2 diabetes (T2D) or oral antidiabetic prescription, active cancer, terminal illness or cognitive impairment, pregnancy, cardiovascular disease, inability to perform moderate-vigorous physical exercise for the next 3 months, major surgery or hospital admission in the last 3 months, haematological disease that interferes with HbA1c determination, presence of any condition (medical, psychological, social or geographical) current or anticipated that limits participation in the study, or participation in another clinical trial will be excluded.

Description of interventions:

The intervention will be designed and implemented by a sports science professional. All groups will perform a minimum of 150 minutes of moderate physical exercise per week or a minimum of 75 minutes of vigorous exercise per week, always performed under the supervision of a sports science professional. During the intervention participants will progress to 300 minutes of moderate physical activity (PA) or 150 of vigorous PA. Prior to the start of the full intervention, participants will undergo a 3-week pre-intervention physical conditioning. Each intervention will last 12 weeks. Before starting the intervention program, participants would be referred to a physician for medical testing and clearance. During all physical exercise sessions, participants will wear a heart rate (HR) device that will relay their HR to a laptop, from which the sports scientist will be able to control the intensity of the session. The heart rate monitor model to be used is the Polar OH1, which has been validated in previous studies. Polar HR monitors have demonstrated a high level of agreement with the electrocardiogram and can therefore be used as a valid measure of HR in both laboratory and field studies to measure HR during moderate-to-vigorous PA (MVPA).

Three exercise modalities will be compared: 1) Aerobic training (AT), 2) AT combined with resistance training (RT) and 3) High intensive interval training (HIIT). During all intervention sessions, participants will wear a HR monitor connected to a computer. In this way, study staff will be able to control the intensity of the session and individualise exercise prescriptions in real time. Heart rate monitoring will be a key element in ensuring that each exercise is performed at the target intensity, by calculating the intensity at which each volunteer performs the exercise based on a percentage of their HR. Despite there are numerous formulas for estimating the maximum heart ratio (HRmax), studies based on meta-analysis reported that [HRmax = 208 - 0.7 × age] is a more reliable option to predict HRmax. Once the HRmax has been estimated, the Karvonen formula will be used to calculate the HR corresponding to a given percentage of intensity, for example, if we want a subject to exercise at 60% of their HRmax, it will be calculated using the Karvonen formula, which takes into account HRmax and basal heart rate (HRB), and is as follows: (HRB + % intensity desired [HRmax - HRB]). This formula has been recommended for both, people with cardiac diseases and athletes due to the accurate characteristics of the formula.

1. Aerobic Training intervention (AT): Perform 50 minutes/day, 3 days/week, totalling 150 min/week at moderate intensity, as recommended by WHO, in a range of 65-75% HRMax. Due to any form of aerobic exercise involving large muscle groups and causes sustained increases in HR is likely to be beneficial, the type of aerobic exercise will be agreed with each group of patients, varying from 4 to 8 people. There will be a choice of exercises and participants will be able to choose a combination of up to 2 different exercises. The participants' choice of the type of activity to be performed is expected to en-courage greater adherence. The range of exercises will be brisk walking or running, swimming, and/or aerobic dancing.
2. Aerobic Training plus Resistance Training intervention (AT+RT): Perform 50 minutes/day, 3 days/week, starting with 50% of 1-repetition maximum (1-RM) and follow a progression of increasing loads up to 75% of 1-RM for optimal gains in strength and insulin action. In each session, between 5 and 10 exercises will be worked on, performing 10-15 repetitions, and progressing to 8-10 lifting as the weight increases, involving the major muscle groups from the core, lower body and upper body. In all sessions there will be a 3-minute warm-up at the beginning of the session and a 2-minute cool-down at the end of the session.
3. High Intensive Interval Training intervention (HIIT): To be considered high intensive the heart rate needs to be above ≥85% . Perform 25 minutes/day, 3 days/week, totalling 75 min/week at a vigorous intensity, as recommended by WHO. Starting with 4 intervals lasting 1 minute keeping in a range of 85-90% HRMax, separated by 1 minute of low intensity activity (no static) (4 × 1 min intervals.) A progression will be followed by increasing the number of circuits, up to 10 (10 × 1 min intervals). In all sessions there will be a 3-minute warm-up at the beginning of the session and a 2-minute cool-down at the end of the session. Although the target population is a sedentary population, we expect the HIIT approach, despite being high intensity, to be well received, due to its growing popularity, as demonstrated by a study in which 62% of inactive participants preferred HIIT to other types of exercise.

Participants in the control group will receive written standard PA recommendations in this phase.

Main dependent variable:

The primary outcome variable is the change in FPG at 15 weeks of follow-up. Secondary dependent variables: glycaemic variability, HbA1c, TG, blood pressure, body composition, waist circumference, transcriptomic biomarkers in blood and quality of life.

Main independent variable The main independent variable is the assigned group.

Statistical analysis Statistical analyses will be performed using R v3.3.1 and Stata v17.0 program. P-values <0.05 will be deemed statistically significant.

* Descriptive analysis, labelling and data cleaning: Assessment of outliers and extreme values, detection and labelling of missing and/or non-applicable values, and description of the distribution of each of the variables. Normality test and scatter plots.
* Descriptive baseline analysis: Sociodemographic characteristics and FPG and continuous blood glucose values by the 3 intervention modalities.
* Main analysis: This will be differentiated for each of the phases and will be done by intention-to-treat and per protocol analysis. A comparison of the decrease in FPG and glycaemic variability between the 3 modalities will be made. The ANOVA test will be used for both phases. If the assumptions of normality are not met, the Kruskal-Wallis test will be applied. A crude analysis, or adjusted for baseline characteristics if necessary, will be performed using general linear models (GLM) to determine the effect of membership in each exercise group on decreasing FPG and glycaemic variability values. A similar analysis will be performed for each of the secondary dependent variables (HbA1c, TG, blood pressure, body composition, waist circumference and quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Overweight (BMI >25 and <35 Kg/m2)
* Inactive (<150 min PA/week)
* With prediabetes (fasting blood glucose 100-126 mg/dl)
* Who have signed the informed consent

Exclusion Criteria:

* People with uncontrolled hypertension
* Diagnosis of T2D or oral anti-diabetic prescription
* Active cancer
* Terminal illness
* Cognitive impairment
* Pregnancy
* Cardiovascular disease
* Inability to perform moderate-vigorous physical exercise for the next 3 months
* Major surgery or hospital admission in the last 3 months
* Haematological disease that interferes with HbA1c determination
* Presence of any condition (medical, psychological, social or geographical) current or anticipated that limits participation in the study
* Participation in another clinical trial will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2023-04-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
fasting plasma glucose | 15 weeks of intervention
  Changes in fasting plasma glucose, revers to normoglycaemia levels

SECONDARY OUTCOMES:
glycaemic variability (measured with continuos glucose monitor: Time in range and MAGE) | 15 weeks of intervention
  improvement in this parameters
HbA1c | 15 weeks of intervention
  improvement in this parameters
transcriptomic biomarkers in blood (PBC) | 15 weeks of intervention
  improvement in this parameters
Triglycerides | 15 weeks of intervention
  improvement in this parameters
Systolic and Diastolic Blood Pressure | 15 weeks of intervention
  improvement in this parameters
body composition (measured by bioimpedance) | 15 weeks of intervention
  improvement in this parameters

CONTACTS AND LOCATIONS:
Overall Officials: Aina Yañez, PhD, Principal Investigator — University of the Balearic Islads (aina.yanez@uib.es)

IPD SHARING:
Plan to Share IPD: No